CLINICAL TRIAL: NCT02374411
Title: A Survey of the Knowledge, Attitudes, and Practice of Surgeons Toward Nutrition Support in HIPEC Patients
Brief Title: Knowledge, Attitudes, and Practice of Surgeons Toward Nutrition Support in HIPEC Patients
Status: Completed | Type: Observational
Sponsor: Edward Hospital (Other)
Responsible Party: Sponsor
Organization: Edward-Elmhurst Health System (Other)
Other Study IDs: EDW091114A
Record Dates: First submitted 2014-09-24; First posted 2015-02-27 (Estimated); Last update posted 2017-02-08 (Estimated); Status verified 2017-02

CONDITIONS: Pseudomyxoma Peritonei; Appendiceal Neoplasms; Pancreatic Neoplasms; Neoplasm Metastasis; Adenocarcinoma; Sarcoma; Uterine Neoplasms
MeSH Terms: conditions — Pseudomyxoma Peritonei; Appendiceal Neoplasms; Pancreatic Neoplasms; Neoplasm Metastasis; Adenocarcinoma; Sarcoma; Uterine Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- HIPEC surgeons

SUMMARY:
The goal of this survey of international HIPEC (Hyperthermic Intraperitoneal Chemotherapy) surgeons is to determine their knowledge of and attitudes towards the nutritional support needs of HIPEC patients and what their practice patterns are with this patient population.

ELIGIBILITY:
Inclusion Criteria:

* Surgeon trained in and performing the HIPEC procedure

Exclusion Criteria:

* Not performing the HIPEC procedure

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: HIPEC surgeons based internationally
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2014-09; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Collect questionnaire data from 150 HIPEC surgeons | Three months
  Questionnaire development was informed by the works of: Karim et al, JPEN 2014 Mar 3, [Epub ahead of print]; Cahill, et al, Critical Care 2014, 18:R96; Vashi et al, Nutrition Journal 2013, 12:118; and Cahill et al, BMC Health Services Research 2014, 14:197.

SECONDARY OUTCOMES:
HIPEC surgeon practices of patient nutritional support assessed by questionnaire | Three months
  Questionnaire development was informed by the works of: Karim et al, JPEN 2014 Mar 3, [Epub ahead of print]; Cahill, et al, Critical Care 2014, 18:R96; Vashi et al, Nutrition Journal 2013, 12:118; and Cahill et al, BMC Health Services Research 2014, 14:197.
HIPEC surgeon attitudes toward patient nutritional support self-assessed by questionnaire | Three months
  Questionnaire development was informed by the works of: Karim et al, JPEN 2014 Mar 3, [Epub ahead of print]; Cahill, et al, Critical Care 2014, 18:R96; Vashi et al, Nutrition Journal 2013, 12:118; and Cahill et al, BMC Health Services Research 2014, 14:197.

CONTACTS AND LOCATIONS:
Overall Officials: George I Salti, MD, Principal Investigator — Edward Hospital
Locations (1):
- Edward Hospital, Naperville, Illinois, United States